CLINICAL TRIAL: NCT03547687
Title: Electrical Stimulation to Reduce Length of Stay and Duration of Intubation in the Neurosciences-intensive Care Unit (NSICU)
Brief Title: Neurosciences-Intensive Care Unit Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michelle Cameron, Associate Professor of Neurology, School of Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018079
Record Dates: First submitted 2018-05-17; First posted 2018-06-06 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Intensive Care (ICU) Myopathy
Keywords: Electrical stimulation; Intubation; ICU discharge
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Electrical Stimulation Treatment (Experimental): Patient will receive electrical stimulation to the quadriceps muscle groups on both lower extremities simultaneously for 45 minutes at a time, for a total of 5 treatments each week (Mon-Sun), for up to 14 days or until ICU discharge, whichever comes first.
  Interventions: Device: Electrical Stimulation Treatment; Device: Neuromuscular Electrical Stimulation Treatment

INTERVENTIONS:
Device: Electrical Stimulation Treatment — An Intelect Neuromuscular Electrical Stimulator (NMES) (Chattanooga Group) device will be used to provide the stimulation. The stimulator will be set up and taken off the patients by a member of the study team or a trained ICU staff member. The stimulation parameters will be as follows:
  Electrode location: Proximal and distal quadriceps Waveform: pulsed biphasic Pulse duration: 300 microseconds Pulse frequency: 35 pulses per second Amplitude: palpable, visible quadriceps muscle contraction On/off time: 5 seconds on, 15 seconds off Ramp up and down time: 2 seconds each
  Other Names: Intelect Neuromuscular Electrical Stimulator (NMES); Intelect Portable Electrotherapy for NMES
Device: Neuromuscular Electrical Stimulation Treatment — If a muscle contraction is not produced with the Intelect NMES portable device, the Vectra Neo Clinical Therapy System (Chattanooga Group) device will be used instead. The stimulator will be set up and taken off the patients by a member of the study team or a trained ICU staff member. The stimulation parameters will be as follows:
  Electrode location: Proximal and distal quadriceps Waveform: pulsed biphasic Pulse duration: 300 microseconds Pulse frequency: 35 pulses per second Amplitude: palpable, visible quadriceps muscle contraction On/off time: 10 seconds on, 30 seconds off Ramp up and down time: 2 seconds each
  Other Names: Vectra Neo Clinical Therapy System

SUMMARY:
Patients admitted to the Neurosciences Intensive Care Unit (NSICU) are at particular risk of developing ICU-associated weakness and myopathy, given the unique risks of early mobilization in these patients, which include increased intracranial pressure, hemodynamic instability, vasospasm, decreased cerebral blood flow with resultant cerebral ischemia, and delirium. Interventions that could provide some of the benefits of early mobilization without these risks would be of great utility in the NSICU. A number of studies have demonstrated that electrical stimulation of the lower extremity muscles, generally the quadriceps, can retard disuse atrophy and loss of strength associated with medical ICU stays, and one study has shown reduced length of intubation and accelerated functional recovery. This pilot trial will evaluate the impact of electrical stimulation on patients in the NSICU, with a hypothesis that electrical stimulation treatments will reduce the length of hospital stay and intubation and improve functional recovery. In this trial, intubated patients admitted to the NSICU will have electrical stimulation applied to the quadriceps muscle groups on both lower extremities simultaneously for 45 minutes at a time for a total of 5 treatments each week, for up to 14 days or until ICU discharge, whichever comes first.

DETAILED DESCRIPTION:
The purpose of this pilot trial is to estimate the effect of electrical stimulation (e-stim) to the bilateral quadriceps on duration of intubation, ICU and hospital length of stay, and functional recovery in the NSICU in comparison to historical matched controls. The objectives of this initial pilot and feasibility study are to estimate the effect size to power a future full scale randomized controlled trial of this intervention and to optimize study logistics for a future full scale trial. The specific aims of the trial are:

Specific Aim 1 - Feasibility: Determine whether at least 4 of 5 planned treatments can be performed as described, and whether there is adequate patient population meeting inclusion criteria available for study

Specific Aim 2 - Efficacy: Evaluate efficacy of e-stim by comparing length of ICU stay (days from admission to "intermediate level of care" ordered in Epic) and duration of intubation (days) of subjects to that of historical controls.

Specific Aim 3 - Exploratory: Evaluate functional recovery (measured by modified Rankin Scale [mRS] and Extended Glasgow Outcome Scale [GOSE] at NSICU discharge) of subjects compared to that of historical controls.

Hypothesis: The investigators hypothesize that e-stim treatments will reduce the length of hospital stay and intubation and improve functional recovery.

The study will be a prospective, feasibility pilot study of 22 subjects enrolled from the NSICU to estimate the effect size to power a future, full scale randomized controlled trial of electrical stimulation. The information learned in the pilot will help the team optimize study logistics for a future full-scale trial. The controls used for comparison will be obtained from an NSICU patient database, using the average values of the outcomes for patients from the previous year who would have met inclusion criteria.

Patients admitted to the NSICU will be screened for eligibility through a review of medical records in Epic by study staff, and approached for consent. Patients with prognosticated prolonged stay will be approached on day 3 to 5 of their ICU stay for enrollment.

For the treatment procedure, electrical stimulation will be applied to the quadriceps muscle groups on both lower extremities simultaneously for 45 minutes at a time. The patient will be positioned either supine or sitting.

An Intelect Neuromuscular Electrical Stimulator (Chattanooga Group) device or an Vectra® Neo Clinical Therapy System device will be used to provide the stimulation. The stimulator will be set up and taken off the patients by a member of the study team or a trained ICU staff member. The stimulation parameters will be as follows:

Electrode location: Proximal and distal quadriceps Waveform: pulsed biphasic Pulse duration: 300 microseconds Pulse frequency: 35 pulses per second Amplitude: palpable, visible quadriceps muscle contraction On/off time: 5 seconds on, 15 seconds off Ramp up and down time: 2 seconds each Total treatment time: 45 ± 15 minutes/day, for a total of 5 treatments each week (Mon-Sun), for up to 14 days or until ICU discharge, whichever comes first.

At NSICU discharge, a member of the study team will assess functional recovery using the modified Rankin Scale (mRS) and the Extended Glasgow Outcome Scale (GOSE). Subjects who withdraw from e-stim treatment may still be assessed with these instruments at discharge, unless they request to withdraw from data collection as well. Subjects may be withdrawn from e-stim treatment without their consent if their physician or the study team decides that it is in their best interest (e.g. due to skin irritation or burns).

All procedures will be performed as part of the research study, and not as standard of care.

Data will be collected from the subjects' medical record in Epic, and from the mRS and GOSE instruments (completed by study staff). All data will be stored in RedCap. Data collected from the medical record will include demographics (sex, age, race), illness information (primary admission diagnosis, severity of critical illness as determined by the Sequential Organ Failure Score (SOFA) and/or APACHE II score), critical illness-associated complications (e.g. deep vein thrombosis, hospital acquired infection, etc.), and medications associated with neuromuscular weakness (e.g. steroids, neuromuscular blockers, etc.).

Analysis plan

Covariates: The following factors may impact outcome, and thus will be collected to assure the groups are comparable:

i. Demographics (sex, age, race) ii. Illness information: primary admission diagnosis, severity of critical illness (Sequential Organ Failure Score (SOFA), APACHE II score) iii. Critical Illness-Associated Complications: complications such as deep vein thrombosis, Hospital-acquired infection, etc. will be recorded as these conditions may impact outcome.

iv. Medications associated with neuromuscular weakness: including but not limited to steroids and neuromuscular blockers

Group Comparisons The study team statistician will analyze the data, and will be blinded to treatment assignment ("Group A" and "Group B", instead of "E-Stim Group" and "Historical Controls"). Descriptive statistics will be used to quantify feasibility. Mean length of stay and mean duration of intubation will be compared between the e-stim group and the historical controls using a t-test. If necessary, a linear regression model for length of stay and/or intubation duration will be used to compare groups while controlling for the potential confounding of covariates. A Wilcoxon rank-sum test will be used to compare the exploratory functional outcome measures between groups, as the mRS and GOSE are both ordinal scales.

The risks involved in the study are all small and mild:

1. Burns - electrical stimulation can cause burns, although this is very rare with the pulsed current that will be used in this study because electricity is only flowing for a very small proportion of the time with this type of current. The risk of burns is also increased if the electrodes have poor contact with the patients' skin. This will be avoided by closely inspecting the electrodes for good contact when applied, by cleaning the skin with water before applying the electrodes, clipping hair in the area of electrodes if present, and by using new electrodes at least weekly, or sooner if they start to adhere poorly.
2. Skin irritation or inflammation - the adhesive on electrical stimulation electrodes, which is similar to tape adhesive, can cause skin irritation in some individuals. Therefore, individuals with tape allergy will be excluded from this study. In addition, if a subject develops skin irritation, the investigators will switch to hypo-allergenic electrodes. If the skin irritation persists, the subject will be withdrawn from the study.
3. Discomfort during the stimulation - if the intensity is high enough an individual may experience discomfort during electrical stimulation. The investigators will limit the stimulation intensity to that sufficient to produce a visible muscle contraction and will discontinue the intervention if the subject either reports pain or has signs of pain e.g. elevated heart rate or blood pressure in response to the stimulation.
4. Delayed muscle soreness - there is a risk of delayed onset muscle soreness in the muscles stimulated. This is similar to the soreness experienced after exercise and will resolve without intervention. This is only likely if the exercise is substantially greater than the individual's usual activity. Although 30 minutes of visible quadriceps contraction is not generally likely to cause delayed onset muscle soreness, it is possible this will occur.
5. There is a small risk of breach of confidentiality.

It is hypothesized but unknown whether there are benefits to e-stim treatment. E-stim may result in reduced duration of hospitalization and intubation, and may improve recovery outcomes.

The devices for this study are the Intelect® Portable Electrotherapy for Neuromuscular Electrical Stimulation and the Vectra® Neo Clinical Therapy System, which are commercially manufactured by Chattanooga. The devices are FDA approved for the prevention of disuse atrophy and also are used for muscle re-education, increasing range of motion, and increasing circulation. These devices are used in commonly in clinical Physical Therapy practice in other patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the NSICU for care for a neurologic illness requiring critical care
* Mechanically ventilated at time of enrollment
* Prognosis for prolonged ICU stay and/or prolonged intubation as evidenced by at least one pre-morbid risk factor: age ≥ 65 years, major medical co-morbidity (ex: heart failure, chronic obstructive pulmonary disease, chronic renal insufficiency, diabetes, poorly controlled hypertension, etc.), or severe acute critical illness (APACHE II >12)

Exclusion Criteria:

* Contraindications to electrical stimulation - demand cardiac pacemaker, implanted cardiac defibrillator, deep brain stimulator, adhesive allergy, pregnancy
* Agitation such that the individual is at risk for pulling off the self-adhesive electrodes
* Moribund prognosis (not expected to survive >48 hours, initiation of comfort measures only)
* Severe peripheral edema
* Receiving vasopressors at the time of enrollment, or hemodynamically unstable
* Severe peripheral neuropathy (ex: acute inflammatory polyneuropathy)
* Receiving paralytic drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cameron, MD, PT, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to the Neuro ICU were screened for eligibility through a review of medical records in Epic by study staff, and approached for consent. Patients with prognosticated prolonged stay were approached on day 2 to 5 of their ICU stay for enrollment. If patients had reversible exclusion criteria, such as hemodynamic instability or elevated intracranial pressures, they were rescreened daily for potential enrollment until day 7.
Groups:
- Electrical Stimulation Treatment: Patient will receive electrical stimulation to the quadriceps muscle groups on both lower extremities simultaneously for 45 minutes at a time, for a total of 5 treatments each week (Mon-Sun), for up to 14 days or until ICU discharge, whichever comes first.
  Electrical Stimulation Treatment: An Intelect Neuromuscular Electrical Stimulator (NMES) (Chattanooga Group) device or a Vectra® Neo Clinical Therapy System will be used to provide the stimulation. The stimulator will be set up and taken off the patients by a member of the study team or a trained ICU staff member. The stimulation parameters will be as follows:
  Electrode location: Proximal and distal quadriceps Waveform: pulsed biphasic Pulse duration: 300-450 microseconds Pulse frequency: 35 pulses per second Amplitude: palpable, visible quadriceps muscle contraction On/off time: 10 seconds on, 30 seconds off Ramp up and down time: 2 seconds each
Period: Overall Study
Arm/Group | Electrical Stimulation Treatment
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Electrical Stimulation Treatment
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (21.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Weight [Mean (Standard Deviation); unit: kilograms] | 74.5 (18.6)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.49 (6.22)
SOFA Score [Mean (Standard Deviation); unit: units on a scale] — Sequential Organ Failure Assessment (SOFA) Score predicts ICU mortality based on patient laboratory values and clinical data. An integer value of 0 to 24 is calculated in the first 24 hours of ICU admission, based on respiratory system, nervous system, cardiovascular system, liver function, coagulation and kidney function. Higher scores correspond to more severe disease and a higher risk of death.
  units on a scale | 6.56 (2.46)
APACHE II Score [Mean (Standard Deviation); unit: units on a scale] — The APACHE II ("Acute Physiology And Chronic Health Evaluation II") is an ICU scoring system to classify severity of disease using patient laboratory values, patients medical comorbidities, and patient clinical characteristics. An integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
  units on a scale | 18.67 (3.57)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Intubation
Description: Duration of intubation in days
Time Frame: Within 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Electrical Stimulation Treatment
Number analyzed (Participants) | 9
days | 10.22 (10.44)

2. Secondary Outcome: Length of Neuroscience Intensive Care Unit Stay
Description: Calculated based on date of admission to Neuroscience Intensive Care Unit (NSICU) and date of transfer from NSICU
Time Frame: Within 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Electrical Stimulation Treatment
Number analyzed (Participants) | 9
days | 13.67 (6.58)

3. Secondary Outcome: Length of Hospital Stay
Description: Calculated based on date of admission to hospital and date of discharge from hospital
Time Frame: Within 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Electrical Stimulation Treatment
Number analyzed (Participants) | 9
days | 29.56 (24.17)

4. Secondary Outcome: Modified Rankin Scale
Description: Modified Rankin Scale at at NSICU transfer, assessed by Nurse Practitioner. Measures degree of disability in patients after neurologic injury. Scale range is 0-6, higher value is a worse outcome.
Time Frame: Within 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Stimulation Treatment
Number analyzed (Participants) | 9
score on a scale | 4.33 (1.73)

5. Secondary Outcome: Glasgow Outcome Scale - Extended
Description: Glasgow Outcome Scale - Extended at NSICU transfer, assessed by Nurse Practitioner. Measures global functional outcomes after neurologic injury. Scale range is 1-8, higher value is a better outcome.
Time Frame: Within 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Stimulation Treatment
Number analyzed (Participants) | 9
score on a scale | 3.44 (2.55)

ADVERSE EVENTS:
Time Frame: Patient was evaluated for adverse events at the time of electrode placement and for 30 minutes after the removal of the electrodes, for a total of 45 minutes with each stimulation treatment for 14 days of treatment or until ICU discharge up to 90 days.
Groups:
- Electrical Stimulation Treatment: Patient will receive electrical stimulation to the quadriceps muscle groups on both lower extremities simultaneously for 45 minutes at a time, for a total of 5 treatments each week (Mon-Sun), for up to 14 days or until ICU discharge, whichever comes first.
  Electrical Stimulation Treatment: An Intelect Neuromuscular Electrical Stimulator (NMES) (Chattanooga Group) device will be used to provide the stimulation. The stimulator will be set up and taken off the patients by a member of the study team or a trained ICU staff member. The stimulation parameters will be as follows:
  Electrode location: Proximal and distal quadriceps Waveform: pulsed biphasic Pulse duration: 300 microseconds Pulse frequency: 35 pulses per second Amplitude: palpable, visible quadriceps muscle contraction On/off time: 5 seconds on, 15 seconds off Ramp up and down time: 2 seconds each
Arm/Group | Electrical Stimulation Treatment
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
We were unable to achieve consistent muscle contraction with the initial portable NMES device. No patients were enrolled for 5 months while another clinical NMES device that had a higher maximum intensity output was obtained. More patients likely qualified than were actually enrolled, as screening and enrollment were limited by study staff availability. Small number of subjects enrolled lead to uninterpretable analysis of historic controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03547687/Prot_SAP_000.pdf